CLINICAL TRIAL: NCT05466409
Title: Training Requirements in Point of Care Ultrasonography of the Upper Airway. A Feasibility Study
Brief Title: Upper Airway Ultrasound Training Requirements
Status: Completed | Type: Observational
Sponsor: University of Ioannina (Other)
Responsible Party: Principal Investigator, Agathi Karakosta, Assistant Professor of Anaesthesiology, University of Ioannina
Other Study IDs: 942
Record Dates: First submitted 2022-07-17; First posted 2022-07-20 (Actual); Last update posted 2022-07-26 (Actual); Status verified 2022-07

CONDITIONS: Airway Management
Keywords: Training; Point-of-care-ultrasound

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Visualization of the hyoid bone — Visualization of the hyoid bone using POCUS of upper airway (probe positioning: transverse plane). Hyoid bone visualization will be assessed as a binary outcome (yes/no).
Other: Visualization of vocal cords — Visualization of the vocal cords through the cricoid cartilage using POCUS of upper airway (probe positioning: transverse plane). Vocal cords visualization will be assessed as a binary outcome (yes/no).
Other: Localization of thyrohyoid membrane — Localization of thyrohyoid membrane using POCUS of upper airway (probe positioning: midsagittal plane). Thyrohyoid membrane visualization will be assessed as a binary outcome (yes/no).
Other: Visualization of epiglottis and pre-epiglottic space — Visualization of epiglottis and pre-epiglottic space using POCUS of upper airway (probe positioning: midsagittal plane). Epiglottis and pre-epiglottic space visualization will be assessed as a binary outcome (yes/no).
Other: Visualization of cricothyroid membrane — Visualization of cricothyroid membrane using POCUS of upper airway (probe positioning: midsagittal plane). Cricothyroid membrane visualization will be assessed as a binary outcome (yes/no).
Other: Visualization of thyroid gland — Visualization of thyroid gland using POCUS of upper airway (probe positioning: transverse plane). Thyroid gland visualization will be assessed as a binary outcome (yes/no).
Other: Hyoid bone to skin distance — Measurement of hyoid bone to skin distance (mm) using POCUS of upper airway (probe positioning: transverse plane).
Other: Anterior commissure to skin distance — Measurement of anterior commissure to skin distance (mm) using POCUS of upper airway (probe positioning: transverse plane).
Other: Epiglottis to skin distance — Measurement of epiglottis to skin distance (mm) using POCUS of upper airway (probe positioning: midsagittal plane).
Other: Thyroid isthmus to skin distance — Measurement of thyroid isthmus to skin distance (mm) using POCUS of upper airway (probe positioning: transverse plane).

SUMMARY:
The applications of point-of-care ultrasonography (POCUS) of the upper airway are growing over the last decade. It's clinical applications include both diagnosis of upper airway pathology as well as pre-intubation airway examination and provision of ultrasound markers of difficult laryngoscopy and/or intubation.

However, it is differentiated from the comprehensive ultrasound examinations traditionally performed by radiologists because it is targeted to answer a specific clinical question in real time. Moreover, ultrasound-guided techniques require knowledge of sonoanatomy and ultrasound operational skills. However, clinicians lack the standardized training that ultrasound technicians and radiologists receive. POCUS training is rarely done in a standardized manner, and even more so, POCUS is rarely conducted under expert's supervision.

The current study investigates the feasibility of upper airway POCUS performed on healthy volunteers by anaesthesia residents using a predefined scanning protocol after attending a structured training course. Assessment of anaesthesia trainees' competence and minimum training requirements were the aim of the study.

DETAILED DESCRIPTION:
Point-of-care (POCUS) of the upper airway has proven a useful tool for airway management as well as diagnosis of upper airway pathology. Although anaesthesiologists are familiar with the use of ultrasound, with peripheral nerve blockade and vascular access representing the most popular applications in anaesthesiology, POCUS is not yet routinely used for airway evaluation. However, the reliability of such examination, which is clinician performed and interpreted, is highly dependent on the operator. Ultrasound-guided techniques require knowledge of sonoanatomy and ultrasound operational skills. Clinicians lack the standardized training that ultrasound technicians and radiologists receive. POCUS training is rarely done in a standardized manner, and even more so, POCUS is rarely conducted under expert's supervision. Insufficient ultrasonographic skills increase the risk of misdiagnosis compromising patient care.

This is a prospective observational study conducted in the University Hospital of Ioannina to investigate the feasibility of upper airway POCUS performed on healthy volunteers by anaesthesia residents using a predefined scanning protocol after attending a structured training course. Assessment of anaesthesia trainees' competence and minimum training requirements are the aim of the study.

All subjects will be healthy volunteer members of the Operating Room (OR) staff. The training course will be shaped in a stepwise manner, beginning with an "education day" that includes a didactic lecture and a hands-on workshop, followed by a "performance week" for competence assessment. During "education day" a predefined scanning protocol will be taught and practiced. An experienced in neck ultrasound radiologist (instructor) will demonstrate the scans and will supervise all trainees. The predefined scanning protocol includes identification of specific structures [(i) visualization of the hyoid bone, (ii) visualization of vocal cords, (iii) localization of thyrohyoid membrane and visualization of epiglottis and pre-epiglottic space, (iv) visualization of cricothyroid membrane, and (v) visualization of thyroid gland)], as well as performance of specific measurements [(i) distance from hyoid bone to skin, (ii) distance from anterior commissure to skin, (iii) distance from epiglottis to skin, and (iv) distance from thyroid isthmus to skin].

During "performance week" all trainees will perform upper airway POCUS to members of the OR staff. The predefined protocol will be applied in each case. A single scan will be allowed for each subject. All subjects will have ultrasound measurements recorded separately by the six trainees and the instructor. The data will be collected at bedside and each participant will be blinded to each other's assessments. Trainees' performance will be assessed by paired calculations of the trainee - instructor differences in all ultrasound measurements of interest.

ELIGIBILITY:
Inclusion Criteria:

- healthy adult volunteers (ASA physical status I and II)

Exclusion Criteria:

* history of congenital or acquired airway abnormalities
* modified Simplified Airway Risk Index (SARI) > 4
* mallampati score > 3
* Body mass index (BMI) > 35 Kg/m2

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy adult volunteers, all members of the Operating Room (OR) staff, not anticipated to have difficult laryngoscopy and/or intubation based on their clinical upper airway evaluation.
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2021-11-29 (Actual); Primary Completion 2021-12-06 (Actual); Study Completion 2021-12-13 (Actual)

PRIMARY OUTCOMES:
T-I differences for hyoid bone to skin distance | 10 days
  Paired calculations of trainee-instructor (T-I) differences (mm) for hyoid bone to skin distance.
T-I differences for anterior commissure to skin distance | 10 days
  Paired calculations of trainee-instructor (T-I) differences (mm) for anterior commissure to skin distance.
T-I differences for epiglottis to skin distance | 10 days
  Paired calculations of trainee-instructor (T-I) differences (mm) for epiglottis to skin distance.
T-I differences for thyroid isthmus to skin distance | 10 days
  Paired calculations of trainee-instructor (T-I) differences (mm) for thyroid isthmus to skin distance.

SECONDARY OUTCOMES:
Hyoid bone visualization | 10 days
  Success rate (%) for hyoid bone visualization using upper airway POCUS (transverse plane).
Vocal cords visualization | 10 days
  Success rate (%) for vocal cords visualization using upper airway POCUS (transverse plane).
Thyrohyoid membrane localization, epiglottis and pre-epiglottic space visualization | 10 days
  Success rate (%) for thyrohyoid membrane localization, epiglottis and pre-epiglottic space visualization using upper airway POCUS. All structures (thyrohyoid membrane, epiglottis and pre-epiglottic space) will be assessed under one view with the probe positioned in the midsagittal plane.
  using upper airway POCUS (transverse plane).
Cricothyroid membrane visualization | 10 days
  Success rate (%) for cricothyroid membrane visualization using upper airway POCUS (midsagittal plane).
Thyroid gland visualization | 10 days
  Success rate (%) for thyroid gland visualization using upper airway POCUS (transverse plane).
Sanning duration | 10 days
  Total duration (seconds) of the predefined scanning protocol.

CONTACTS AND LOCATIONS:
Locations (1):
- Univesity Hospital of Ioannina, Ioannina, Epirus, Greece

IPD SHARING:
Plan to Share IPD: Undecided